CLINICAL TRIAL: NCT04260802
Title: A Phase 1b/2a Two-Part, Open-Label, Multicenter Study to Evaluate the Safety and Pharmacokinetics of OC-001 as Monotherapy and in Combination With an Anti-PD-1/Anti-PD-L1 Antibody in Patients With Selected Locally Advanced or Metastatic Cancers
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of OC-001 in Patients With Locally Advanced or Metastatic Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Ocellaris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCEL-01
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Neoplasms; Metastatic Cancer; Triple Negative Breast Cancer; Gastric Cancer; Cervical Cancer; Ovarian Cancer; Hepatocellular Carcinoma; Squamous Cell Carcinoma of Head and Neck; Urothelial Carcinoma; Urothelial Neoplasm; Non Small Cell Lung Cancer; Renal Cell Carcinoma; Locally Advanced Solid Tumor; Locally Advanced Malignant Neoplasm; Squamous Cell Carcinoma; Sarcoma; Merkel Cell Carcinoma; Bladder Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Stomach Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Squamous Cell; Sarcoma; Carcinoma, Merkel Cell; Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug: Phase 1b: Dose Escalation (monotherapy) (Experimental): Escalating doses of OC-001 administered intravenously (IV)
- Drug: Phase 1b Dose: Escalation (Combination therapy) (Experimental): Escalating doses of OC-001 administered by IV in combination Avelumab.
  Interventions: Drug: Drug: OC-001 in Combination with Avelumab
- Drug: Phase 2a (Experimental): Doses of OC-001 administered by IV in combination with Avelumab b)
  Interventions: Drug: Drug: OC-001 in Combination with Avelumab

INTERVENTIONS:
Drug: OC-001 — Administered IV.
Drug: Drug: OC-001 in Combination with Avelumab — Administered IV.
  Arms: Drug: Phase 1b Dose: Escalation (Combination therapy); Drug: Phase 2a

SUMMARY:
This study will investigate OC-001 as monotherapy, and in combination with, Avelumab, in various cancer types

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. Have histological or cytological evidence of a diagnosis of selected cancer types that is locally advanced and/or metastatic

1. Have the presence of evaluable disease for the Phase 1b Monotherapy
2. Have the presence of evaluable and measurable disease for the Phase 1b combination part and the Phase 2a part of the study.
3. The patient must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have failed to provide clinical benefit for their disease or patients who have refused standard treatments.

   2. Cancer treatment and type criteria:
   * Have received at least 1 but no more than 4 prior systemic therapies for locally advanced or metastatic disease (e.g., hormonal, cytotoxic, etc.) for the following cancer types, for Phase 1b:
   * Triple Negative Breast Cancer (TNBC): Must have recurrent/refractory TNBC, defined as any breast cancer that expresses less than (˂)1% estrogen receptor (ER), ˂ 1% progesterone receptor (PR), and is Human Epidermal Growth Factor Receptor 2 (Her2) negative. Must have failed at least one chemotherapy regimen.
   * Gastric Cancer: Must have failed a platinum-containing chemotherapy regime.
   * Cervical Cancer: Must have failed at least one chemotherapy regimen.
   * Ovarian Cancer: Must have failed a platinum-containing chemotherapy regimen but not be platinum refractory.
   * Hepatocellular Cell Carcinoma (HCC): May have failed unlimited liver local therapies.
   * Sarcoma: Must have failed at least one prior chemotherapy regimen.
   * Squamous Cell Carcinoma of Head and Neck (SCCHN): Must have failed a platinum-containing chemotherapy regiment. Must have failed a previous immune checkpoint inhibitor.
   * Bladder Cancer: Must have failed a platinum-containing chemotherapy regiment. Must have failed a previous immune checkpoint inhibitor.
   * Non Small Cell Lung Cancer (NSCLC): Must have failed a platinum-containing chemotherapy regimen or Immuno Oncology (IO) agent in the first line. Must have failed a previous immune checkpoint inhibitor. Must not have any history of tumors that test positive for epidermal growth factor receptor (EGFR), Receptor Tyrosine Kinase (ROS1), Anaplastic Lymphoma Kinase (ALK) mutations or ALK fusions or any other mutations for which tyrosine kinase inhibitors are available.
   * Renal Cell Carcinoma (RCC): Must have failed at least one prior systemic therapy. Must have failed a previous IO agent.
   * Urothelial Cancer: Must have failed at least one prior systemic therapy. Must have failed a previous IO agent.
   * Merkel Cell: Must have failed at least 1 prior systemic therapy for advanced disease and may have failed a previous IO agent.
   * Squamous Cell Carcinoma of the Skin: Must have failed at least 1 prior systemic therapy for advanced disease and may have failed a previous IO agent.

     3. Phase 1b - combination dose escalation:
   * Cervical Cancer Must have failed at least 1 chemotherapy regimen.
   * Bladder Cancer Must have failed a platinum-containing chemotherapy regimen. Must have failed a previous immune checkpoint inhibitor.
   * RCC Must have failed at least 1 prior systemic therapy. Must have failed a previous IO agent.
   * Urothelial cancer Must have failed at least 1 prior systemic therapy. Must have failed a previous IO agent.
   * Diffuse large B cell lymphoma Must have failed prior rituximab therapy. May have failed prior chemotherapy or other IO agents.
   * NSCLC Must have failed a single agent PD-1 or PD-L1 inhibitor as the last regimen and must have responded to the agent.
   * Must not have any history of tumors that test positive for EGFR, ROS1, ALK mutations or ALK fusions, or any other mutations for which tyrosine kinase inhibitors are available or are under development.

     4. For Phase 2a: Must have histological or cytological confirmation of a solid tumor that is locally advanced or metastatic. At least two cancer type will be selected amongst the ones evaluated in the Phase 1b combination dose escalation part of the study.

     5. Have adequate organ function 6 Have a performance status (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale 7 Have discontinued cytotoxic therapy, biologic therapy, immunotherapy, radiotherapy, and cancer-related hormonal therapy at least 21 days prior to study enrollment 8. Are recovered or recovering from the acute adverse effects of any chemotherapy, biologic, therapy, immunotherapy, cancer-related hormonal therapy, or radiotherapy 9. Patients who have had major surgery must be fully recovered and greater than (≥)4 weeks post-operative 10. Men with partners of child-bearing potential or women with child-bearing potential must agree to use a medically approved contraceptive method during and for at least 12 weeks following the last dose of study drug (e.g., intrauterine device (IUD), birth control pills, or barrier method) 11. Women of child-bearing potential must have a negative serum pregnancy test documented 12. Have an estimated life expectancy of at least 3 months

   Exclusion Criteria:
   1. Have symptomatic central nervous system (CNS) metastasis. Patients with treated CNS metastases are eligible for this study if they are asymptomatic and off of corticosteroids for a minimum of 7 days. Patients with primary brain tumors are not eligible
   2. Have a history of major organ transplant (e.g., heart, lungs, liver, and kidney) or an autologous or allogeneic hematopoietic stem cell transplant
   3. Females who are pregnant or nursing
   4. Have known, symptomatic acquired immuno deficiency syndrome (AIDS) or active hepatitis A, B or C
   5. Previous treatment-related, severe (≥Grade 3) Adverse Event (AE) or any neurologic or ocular AE while receiving an IO agent
   6. Active or prior documented autoimmune disease within the past 2 years Patients with vitiligo, Grave's disease or psoriasis not requiring systemic treatment within the past 2 years are eligible
   7. Active or prior documented inflammatory bowel disease
   8. History of tuberculosis, interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required corticosteroid therapy
   9. Receipt of live attenuated vaccination within 28 days prior
   10. Current or prior use of immunosuppressive medication within 28 days prior
   11. Are currently enrolled in another clinical study of an investigational medicinal product
   12. Have a second primary malignancy that may affect the interpretation of results
   13. Are unwilling or unable to participate in, or do not have tissue adequate for a tumor biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with a Dose Limiting Toxicity (DLT) in Phase 1b | Baseline through Cycle 1 (Day 28)
  A Dose-Limiting Toxicity (DLT) is defined as an Adverse Event (AE) that is likely related to the study medication or combination, and fulfills any one of the criteria identified in the Common Terminology Criteria for Adverse Events (CTCAE, Version 5)
Number of participants with any Serious Adverse Event or Treatment-Emergent Adverse Event in Phase 2a | Baseline up to two years
  Number of participants with any Serious Adverse Event or Treatment-Emergent Adverse Event in Phase 2a

SECONDARY OUTCOMES:
Area Under the OC-001 Plasma Concentration Time Curve (AUC) in Phase 1b | Baseline through 12 weeks
  After single and multiple dose administration
Maximum Observed OC-001 Concentration (Cmax) in Phase 1b | Baseline through 12 weeks
  After single and multiple dose administration
Time to reach OC-001 Cmax (Tmax) in Phase 1b | Baseline through 12 weeks
  Time of maximum concentration observed
Minimum Observed OC-001 Concentration (Cmin) in Phase 1b | Baseline through 12 weeks
  After single and multiple dose administration
Overall Response Rate (ORR) in Phase 2a | Baseline up to two years
  In combination with Avelumab
Progression Free Survival (PFS) in Phase 2a | Baseline up to two years
  In combination with Avelumab
Duration of Response (DOR) in Phase 2a | Baseline up to two years
  In combination with Avelumab
Time to Response (TTR) in Phase 2a | Baseline up to two years
  In combination with Avelumab
Disease Control Rate (DCR) in Phase 2a | Baseline up to two years
  In combination with Avelumab
Overall Survival (OS) in Phase 2a | Baseline up to two years
  In combination with Avelumab
One-Year Survival Rate in Phase 2a | Baseline up to two years
  In combination with Avelumab
Maximum Observed OC-001 Concentration (Cmax) in Phase 2a | Baseline through 12 weeks
  In combination with Avelumab
Minimum Observed OC-001 Concentration (Cmin) in Phase 2a | Baseline through 12 weeks
  In combination with Avelumab
Trough drug concentration of OC-001 (Ctrough) in Phase 2a | Baseline through 12 weeks
  In combination with Avelumab

CONTACTS AND LOCATIONS:
Overall Officials: Ocellaris Pharma, Inc, Study Director — Ocellaris Pharma, Inc.
Locations (5):
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Hospital Cancer Centre (OHRI), Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital - Clinical Research Unit, Montreal, Quebec